CLINICAL TRIAL: NCT02880176
Title: Steps to Eliminate Postoperative Problems
Acronym: STEPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 825215; UL1TR000003 (NIH)
Record Dates: First submitted 2016-08-17; First posted 2016-08-26 (Estimated); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Bladder Cancer
Keywords: Behavioral Economics; Financial Incentives; Bladder Cancer; Ambulation; Surgical Co-Morbidity; Fitbit; Mobile Health; Radical Cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Financial Incentive (Experimental): Financial Incentive to Increase Ambulation: A financial reward is given on a per day basis when subject meets daily step goal, 1/5 chance to win additional monetary prize if patient uploads step count data for at least 75% of study days.
  Subjects will use Fitbit Zip to track step counts
  Interventions: Other: Financial Incentive to Increase Ambulation
- Control (Education) (No Intervention): Subjects in this group will receive standard education on the benefits of post-surgery ambulation only Subjects will use Fitbit Zips to track step counts

INTERVENTIONS:
Other: Financial Incentive to Increase Ambulation — Financial Incentive and possibility for financial lottery entry in addition to education on the benefits of post-surgery ambulation
  Arms: Financial Incentive

SUMMARY:
Radical cystectomy with urinary diversion is associated with substantial perioperative morbidity, including deep venous thrombosis, prolonged ileus, and postoperative functional decline. Post-operative morbidity after cystectomy prolongs the length of stay, increases the risk of readmission, and adds substantially to health care costs. Protocols that emphasize early and frequent ambulation after surgery decreases post-operative morbidity, but poor patient adherence diminishes the effectiveness of these protocols, which are currently implemented only during the hospital stay. Financial incentives overcome present bias and offer a novel and practical approach to increasing ambulation during the post-operative period in the hospital and also after discharge. This application proposes a pilot randomized, controlled trial to estimate the effect size of financial incentives on achieving a patient-specific daily step goal in the hospital and post-discharge for 1 month following radical cystectomy. Secondary outcomes include step count, composite morbidity, and functional decline. Forty-six adults with bladder cancer undergoing radical cystectomy at the Hospital of the University of Pennsylvania will be randomized to either control (education of step goal with monitoring and daily feedback) or a gain financial incentive combined with a lottery incentive if they achieve 75% of the daily goals during the study period. Fitbit Zips will be used to measure step counts for all participants. This proposal will provide the preliminary data needed to design future, larger trials that will test the effect of financial incentives to increase ambulation on post operative complications, readmissions, and functional decline.

DETAILED DESCRIPTION:
In this application, a randomized controlled trial will be used to test the hypothesis that small financial incentives can be used to increase post-operative ambulation. The randomized controlled trial design is necessary to demonstrate a causal relationship between the intervention (provision of financial incentives)and the outcome (increased ambulation). This design will also provide preliminary data (e.g. effect sizes, feasibility) needed to design larger trials that will determine whether increases in ambulation produced by financial incentives can be translated into decreases in clinically relevant outcomes such as post-operative complications, readmissions, and functional decline in patients undergoing major abdominal surgery.

All participants will receive education about the importance of early ambulation and knowledge of their daily step goals. A Fitbit Zip, a commercially available activity tracking device with the ability to record and wirelessly upload step counts, will be provided to each participant to measure the outcome of daily step counts for a lead in period of 1-2 weeks before surgery and 30 days after surgery with the option for patients to continue to submit data independently for up to 90 days after surgery. The lead-in period will provide data to determine a patient-specific daily step count baseline. Step count goals will change each week and be determined by a set-percentage of the patient-specific baseline. The percentages will be as follows: 10% of baseline for week 1, 25% of baseline for week 2, 40% of baseline for week 3, and 55% of baseline for week 4. Data will be collected using the Way To Health platform, a digital platform specifically designed to facilitate randomized controlled trials testing interventions increase health promoting behavior.

Participants will be randomized using simple balanced randomization into one of two arms: "control" or "financial incentives". Individuals will be informed if they fail to achieve adequate steps and would have otherwise been eligible for payments in order to leverage regret aversion. The financial incentive is framed as a "gain" rather than a "loss" because striving to achieve a positive reward may provide the necessary support to positively motivate patients who just had major, painful surgery. Small definite payments are combined with larger lottery-based payments to provide ongoing feedback coupled with the possibility of winning a higher magnitude reward. Automated notification about payments will be delivered through the participant's preferred mode of communication (e.g., phone call, email). Patients will track their earnings and step count over time through Way to Health.

Beginning shortly before the planned surgery and continuing for 30 days after date of surgery, all participants will use Fitbit Zips to measure daily step counts. Patients will have the option of submitting up to 90 days of post-operative data. Post-operative ambulation has been repeatedly demonstrated to be beneficial to recovery by a number of different metrics, and the Zip device has been shown to be an accurate measure of step counts. The Stanford Health Assessment Questionnaire (SHAQ) is a broadly used and validated questionnaire which, in its shortened form, assesses subjects ability to perform 20 different actions and the need for assistance with these actions. It also captures patients global assessments of pain and well-being. This will be administered preoperatively, 30 days post-operatively, and 90 days postoperatively to measured post-operative functional decline. The International Physical Activity Questionnaire (IPAQ) Short Seven Day form quantifies patient reported levels of physical activity over the seven days prior to the interview. It is similarly broadly used and has been previously validated against accelerometer data. This will be administered preoperatively, 30 days post-operatively, and 90 days postoperatively to measure post-operative decline in physical activity and to discover differences in baseline physical activity that are not captured by preoperative step-count data.The Multidimensional Scale of Perceived Social Support (MPPSS) is a validated tool for assessing patient's self-assessed degree of support from others. Prior research has suggested social support as an important factor in exercise behavior, which is consistent with our clinical observations. This will be administered pre-operatively and a 30 and 90 days post-operatively to help account for confounding by this important and otherwise unmeasured variable.

ELIGIBILITY:
Inclusion Criteria:

* Planning to undergo radical cystectomy (either with ileal conduit, Indiana pouch, neobladder (e.g., Studer or Hautmann pouch) at the University of Pennsylvania
* Patient has been diagnosed with bladder cancer
* Patient is at least 21 years of age
* Patient is ambulatory with baseline ECOG performance status less than or equal to 2

Exclusion Criteria:

* Patient knows he or she will be unable or unwilling to use a mobile device and online tool to upload activity data
* Poor preoperative performance status (ECOG 3 or greater)
* Plan for cystectomy without cutaneous ureterostomies (without a bowel diversion)
* Non-English speakers
* Patient is non-ambulatory
* Patient is incapable of consenting himself or herself prior to surgery (Because participating in this trial involves ongoing effort on the part of the subject, patients who are incapable of consenting for themselves at baseline are excluded)
* Patients who do not have at least 24 hours of pre-operation ambulation data

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-08; Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Tasian, MD,MSc,MSCE, Principal Investigator — Children's Hospital of Philadelphia; Thomas Guzzo, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stimson CJ, Chang SS, Barocas DA, Humphrey JE, Patel SG, Clark PE, Smith JA Jr, Cookson MS. Early and late perioperative outcomes following radical cystectomy: 90-day readmissions, morbidity and mortality in a contemporary series. J Urol. 2010 Oct;184(4):1296-300. doi: 10.1016/j.juro.2010.06.007. Epub 2010 Aug 17. PMID 20723939
- [Background] Gandaglia G, Varda B, Sood A, Pucheril D, Konijeti R, Sammon JD, Sukumar S, Menon M, Sun M, Chang SL, Montorsi F, Kibel AS, Trinh QD. Short-term perioperative outcomes of patients treated with radical cystectomy for bladder cancer included in the National Surgical Quality Improvement Program (NSQIP) database. Can Urol Assoc J. 2014 Sep;8(9-10):E681-7. doi: 10.5489/cuaj.2069. PMID 25408807
- [Background] Tan HJ, Kaplan AL, Chuang RJ, Kwan L, Filson CP, Litwin MS. The Cost Burden of Complications after Major Surgery for Urological Cancer: Opportunities for Value Creation in Urology. Urol Pract. 2016 Mar;3(2):81-89. doi: 10.1016/j.urpr.2015.05.002. Epub 2015 Dec 29. PMID 37592482
- [Background] Pashikanti L, Von Ah D. Impact of early mobilization protocol on the medical-surgical inpatient population: an integrated review of literature. Clin Nurse Spec. 2012 Mar-Apr;26(2):87-94. doi: 10.1097/NUR.0b013e31824590e6. PMID 22336934
- [Background] Raue W, Haase O, Junghans T, Scharfenberg M, Muller JM, Schwenk W. 'Fast-track' multimodal rehabilitation program improves outcome after laparoscopic sigmoidectomy: a controlled prospective evaluation. Surg Endosc. 2004 Oct;18(10):1463-8. doi: 10.1007/s00464-003-9238-y. Epub 2004 Aug 26. PMID 15791370
- [Background] Padula CA, Hughes C, Baumhover L. Impact of a nurse-driven mobility protocol on functional decline in hospitalized older adults. J Nurs Care Qual. 2009 Oct-Dec;24(4):325-31. doi: 10.1097/NCQ.0b013e3181a4f79b. PMID 19395979
- [Background] Baird G, Maxson P, Wrobleski D, Luna BS. Fast-track colorectal surgery program reduces hospital length of stay. Clin Nurse Spec. 2010 Jul-Aug;24(4):202-8. doi: 10.1097/NUR.0b013e3181e3604c. PMID 20526121
- [Background] Gustafsson UO, Hausel J, Thorell A, Ljungqvist O, Soop M, Nygren J; Enhanced Recovery After Surgery Study Group. Adherence to the enhanced recovery after surgery protocol and outcomes after colorectal cancer surgery. Arch Surg. 2011 May;146(5):571-7. doi: 10.1001/archsurg.2010.309. Epub 2011 Jan 17. PMID 21242424
- [Background] Lee TG, Kang SB, Kim DW, Hong S, Heo SC, Park KJ. Comparison of early mobilization and diet rehabilitation program with conventional care after laparoscopic colon surgery: a prospective randomized controlled trial. Dis Colon Rectum. 2011 Jan;54(1):21-8. doi: 10.1007/DCR.0b013e3181fcdb3e. PMID 21160309
- [Background] Kibler VA, Hayes RM, Johnson DE, Anderson LW, Just SL, Wells NL. Cultivating quality: early postoperative ambulation: back to basics. Am J Nurs. 2012 Apr;112(4):63-9. doi: 10.1097/01.NAJ.0000413460.45487.ea. No abstract available. PMID 22456575
- [Background] Loewenstein G, Brennan T, Volpp KG. Asymmetric paternalism to improve health behaviors. JAMA. 2007 Nov 28;298(20):2415-7. doi: 10.1001/jama.298.20.2415. No abstract available. PMID 18042920
- [Background] Haisley E, Volpp KG, Pellathy T, Loewenstein G. The impact of alternative incentive schemes on completion of health risk assessments. Am J Health Promot. 2012 Jan-Feb;26(3):184-8. doi: 10.4278/ajhp.100729-ARB-257. PMID 22208418
- [Background] Strully KW, Fowler JH, Murabito JM, Benjamin EJ, Levy D, Christakis NA. Aspirin use and cardiovascular events in social networks. Soc Sci Med. 2012 Apr;74(7):1125-9. doi: 10.1016/j.socscimed.2011.12.033. Epub 2012 Feb 4. PMID 22361089
- [Background] Christakis NA, Fowler JH. The spread of obesity in a large social network over 32 years. N Engl J Med. 2007 Jul 26;357(4):370-9. doi: 10.1056/NEJMsa066082. Epub 2007 Jul 25. PMID 17652652
- [Background] Thaler R, Sunstein C. Nudge: improving decisions about health, wealth and happiness. New Haven, CT: Yale University Press; 2008.
- [Background] Volpp KG, Gurmankin Levy A, Asch DA, Berlin JA, Murphy JJ, Gomez A, Sox H, Zhu J, Lerman C. A randomized controlled trial of financial incentives for smoking cessation. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):12-8. doi: 10.1158/1055-9965.EPI-05-0314. PMID 16434580
- [Background] Volpp KG, Loewenstein G, Troxel AB, Doshi J, Price M, Laskin M, Kimmel SE. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res. 2008 Dec 23;8:272. doi: 10.1186/1472-6963-8-272. PMID 19102784
- [Background] Volpp KG, Troxel AB, Pauly MV, Glick HA, Puig A, Asch DA, Galvin R, Zhu J, Wan F, DeGuzman J, Corbett E, Weiner J, Audrain-McGovern J. A randomized, controlled trial of financial incentives for smoking cessation. N Engl J Med. 2009 Feb 12;360(7):699-709. doi: 10.1056/NEJMsa0806819. PMID 19213683
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Loewenstein G, Asch DA, Volpp KG. Behavioral economics holds potential to deliver better results for patients, insurers, and employers. Health Aff (Millwood). 2013 Jul;32(7):1244-50. doi: 10.1377/hlthaff.2012.1163. PMID 23836740
- [Background] John LK, Loewenstein G, Troxel AB, Norton L, Fassbender JE, Volpp KG. Financial incentives for extended weight loss: a randomized, controlled trial. J Gen Intern Med. 2011 Jun;26(6):621-6. doi: 10.1007/s11606-010-1628-y. Epub 2011 Jan 20. PMID 21249462
- [Background] Long JA, Jahnle EC, Richardson DM, Loewenstein G, Volpp KG. Peer mentoring and financial incentives to improve glucose control in African American veterans: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):416-24. doi: 10.7326/0003-4819-156-6-201203200-00004. PMID 22431674
- [Background] Turner BJ, Hollenbeak CS, Liang Y, Pandit K, Joseph S, Weiner MG. A randomized trial of peer coach and office staff support to reduce coronary heart disease risk in African-Americans with uncontrolled hypertension. J Gen Intern Med. 2012 Oct;27(10):1258-64. doi: 10.1007/s11606-012-2095-4. Epub 2012 May 9. PMID 22570108
- [Background] Kullgren JT, Troxel AB, Loewenstein G, Asch DA, Norton LA, Wesby L, Tao Y, Zhu J, Volpp KG. Individual- versus group-based financial incentives for weight loss: a randomized, controlled trial. Ann Intern Med. 2013 Apr 2;158(7):505-14. doi: 10.7326/0003-4819-158-7-201304020-00002. PMID 23546562
- [Background] Jeffery RW, Forster JL, Snell MK. Promoting weight control at the worksite: a pilot program of self-motivation using payroll-based incentives. Prev Med. 1985 Mar;14(2):187-94. doi: 10.1016/0091-7435(85)90034-9. PMID 4048081
- [Background] Forster JL, Jeffery RW, Sullivan S, Snell MK. A work-site weight control program using financial incentives collected through payroll deduction. J Occup Med. 1985 Nov;27(11):804-8. doi: 10.1097/00043764-198511000-00011. PMID 4067685
- [Background] Petry NM, Alessi SM, Marx J, Austin M, Tardif M. Vouchers versus prizes: contingency management treatment of substance abusers in community settings. J Consult Clin Psychol. 2005 Dec;73(6):1005-14. doi: 10.1037/0022-006X.73.6.1005. PMID 16392974
- [Background] Heisler M. Different models to mobilize peer support to improve diabetes self-management and clinical outcomes: evidence, logistics, evaluation considerations and needs for future research. Fam Pract. 2010 Jun;27 Suppl 1(Suppl 1):i23-32. doi: 10.1093/fampra/cmp003. Epub 2009 Mar 17. PMID 19293400 (Retraction: PMID 22850799 Fam Pract. 2012 Aug;29(4):497)
- [Background] Sallis R, Roddy-Sturm Y, Chijioke E, Litman K, Kanter MH, Huang BZ, Shen E, Nguyen HQ. Stepping toward discharge: Level of ambulation in hospitalized patients. J Hosp Med. 2015 Jun;10(6):384-9. doi: 10.1002/jhm.2343. Epub 2015 Mar 9. PMID 25755217
- [Background] Patel MS, Asch DA, Rosin R, Small DS, Bellamy SL, Heuer J, Sproat S, Hyson C, Haff N, Lee SM, Wesby L, Hoffer K, Shuttleworth D, Taylor DH, Hilbert V, Zhu J, Yang L, Wang X, Volpp KG. Framing Financial Incentives to Increase Physical Activity Among Overweight and Obese Adults: A Randomized, Controlled Trial. Ann Intern Med. 2016 Mar 15;164(6):385-94. doi: 10.7326/M15-1635. Epub 2016 Feb 16. PMID 26881417
- [Background] Case MA, Burwick HA, Volpp KG, Patel MS. Accuracy of smartphone applications and wearable devices for tracking physical activity data. JAMA. 2015 Feb 10;313(6):625-6. doi: 10.1001/jama.2014.17841. No abstract available. PMID 25668268
- [Background] Parker SJ, Jessel S, Richardson JE, Reid MC. Older adults are mobile too!Identifying the barriers and facilitators to older adults' use of mHealth for pain management. BMC Geriatr. 2013 May 6;13:43. doi: 10.1186/1471-2318-13-43. PMID 23647949
- [Background] Kwon S, Symons R, Yukawa M, Dasher N, Legner V, Flum DR. Evaluating the association of preoperative functional status and postoperative functional decline in older patients undergoing major surgery. Am Surg. 2012 Dec;78(12):1336-44. PMID 23265122
- [Background] Fries JF, Spitz P, Kraines RG, Holman HR. Measurement of patient outcome in arthritis. Arthritis Rheum. 1980 Feb;23(2):137-45. doi: 10.1002/art.1780230202. PMID 7362664
- [Background] Sen AP, Sewell TB, Riley EB, Stearman B, Bellamy SL, Hu MF, Tao Y, Zhu J, Park JD, Loewenstein G, Asch DA, Volpp KG. Financial incentives for home-based health monitoring: a randomized controlled trial. J Gen Intern Med. 2014 May;29(5):770-7. doi: 10.1007/s11606-014-2778-0. Epub 2014 Feb 13. PMID 24522623
- [Background] Mavros MN, Athanasiou S, Gkegkes ID, Polyzos KA, Peppas G, Falagas ME. Do psychological variables affect early surgical recovery? PLoS One. 2011;6(5):e20306. doi: 10.1371/journal.pone.0020306. Epub 2011 May 25. PMID 21633506
- [Background] Bruce B, Fries JF. The Stanford Health Assessment Questionnaire: dimensions and practical applications. Health Qual Life Outcomes. 2003 Jun 9;1:20. doi: 10.1186/1477-7525-1-20. PMID 12831398
- [Background] Fogelholm M, Malmberg J, Suni J, Santtila M, Kyrolainen H, Mantysaari M, Oja P. International Physical Activity Questionnaire: Validity against fitness. Med Sci Sports Exerc. 2006 Apr;38(4):753-60. doi: 10.1249/01.mss.0000194075.16960.20. PMID 16679993
- [Background] Bagherian-Sararoudi R, Hajian A, Ehsan HB, Sarafraz MR, Zimet GD. Psychometric properties of the persian version of the multidimensional scale of perceived social support in iran. Int J Prev Med. 2013 Nov;4(11):1277-81. PMID 24404362
- [Background] Oka RK, King AC, Young DR. Sources of social support as predictors of exercise adherence in women and men ages 50 to 65 years. Womens Health. 1995 Summer;1(2):161-75. PMID 9373378
- [Background] Brown CJ, Williams BR, Woodby LL, Davis LL, Allman RM. Barriers to mobility during hospitalization from the perspectives of older patients and their nurses and physicians. J Hosp Med. 2007 Sep;2(5):305-13. doi: 10.1002/jhm.209. PMID 17935241
- [Background] Fisher SR, Graham JE, Brown CJ, Galloway RV, Ottenbacher KJ, Allman RM, Ostir GV. Factors that differentiate level of ambulation in hospitalised older adults. Age Ageing. 2012 Jan;41(1):107-11. doi: 10.1093/ageing/afr110. Epub 2011 Sep 9. No abstract available. PMID 21908470
- [Background] Agostini PJ, Naidu B, Rajesh P, Steyn R, Bishay E, Kalkat M, Singh S. Potentially modifiable factors contribute to limitation in physical activity following thoracotomy and lung resection: a prospective observational study. J Cardiothorac Surg. 2014 Sep 27;9:128. doi: 10.1186/1749-8090-9-128. PMID 25262229
- [Background] Fisher SR, Kuo YF, Graham JE, Ottenbacher KJ, Ostir GV. Early ambulation and length of stay in older adults hospitalized for acute illness. Arch Intern Med. 2010 Nov 22;170(21):1942-3. doi: 10.1001/archinternmed.2010.422. No abstract available. PMID 21098357
- [Background] Magheli A, Knoll N, Lein M, Hinz S, Kempkensteffen C, Gralla O. Impact of fast-track postoperative care on intestinal function, pain, and length of hospital stay after laparoscopic radical prostatectomy. J Endourol. 2011 Jul;25(7):1143-7. doi: 10.1089/end.2011.0020. PMID 21740262

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Exceeded recruitment goal.
Period: Overall Study
Arm/Group | Financial Incentive | Control (Education)
Started | 23 | 11
Underwent Cystectomy | 22 | 11
Collected Postop Step Data | 22 | 11
Responded to 30 Day Survey | 20 | 9
Completed | 20 | 9
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Financial Incentive | Control (Education) | Total
Number analyzed (Participants) | 22 | 11 | 33
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.5 [62 to 72] | 65 [62 to 72] | 65 [60 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 21 | 9 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Step Goal Completed
Description: Number of days during the study period that each subject reaches their step goal
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Financial Incentive | Control (Education)
Number analyzed (Participants) | 22 | 11
days | 4.5 [0 to 16] | 9 [6 to 15]

2. Secondary Outcome: Number of Steps Taken Per Day
Description: Average number of steps taken per day in the 30 day postoperative period. Note that the average number of steps taken per day is calculated separately for each patient as simply (total number of steps taken in the 30 day postoperative period)/30. For the purposes of comparing the two study groups, nonparametric tests and medians are used. Thus the "measure type" listed in the "Outcome Measure Data Table" is correctly listed as "median". For example, in the Financial Incentive arm, we report a median average number of steps per day as 979, implying that half of the patients walked fewer than 979 steps on an average day and half of the patients walked more than 979 steps on an average day in that group.
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: steps per day
Arm/Group | Financial Incentive | Control (Education)
Number analyzed (Participants) | 22 | 11
steps per day | 979 [505 to 2646] | 1191 [788 to 1846]

3. Secondary Outcome: Composite Morbidity Outcome of Complications, Unplanned Readmissions, or Emergency Department Visits
Description: Binary variable reflecting whether or not patient suffered any of the following: any postoperative complication, any unplanned readmission, any presentation to the emergency department within 30 days after surgery.
Time Frame: 30 days
Population: Protocol revised to remove this outcome. No data collected.
Arm/Group | Financial Incentive | Control (Education)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Functional Decline as Assessed by the Stanford Health Assessment Questionnaire (SHAQ)
Description: 30-day postoperative Stanford Health Assessment Questionnaire Disability Index (SHAQ) score, indicating subjects ability to perform daily tasks.
  Scores range continuously from 0-4 representing no disability to complete disability respectively. Scores >2 are usually considered severe disability.
  The total score is computed as the mean of 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Each category consists of a list of 2-3 actions. The participant selects whether they are able to perform each action "without any difficulty", "with some difficulty", "with much difficulty", or "unable to do". These selections are scored 0-4 respectively. The category is assigned the maximum score of its component actions. If the subject requires assistance from a person or device for an individual action, the minimum score for that action is 2.
Time Frame: 1 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Financial Incentive | Control (Education)
Number analyzed (Participants) | 20 | 9
units on a scale | 1.25 [1.0 to 1.5] | 1.38 [1.1 to 1.8]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Financial Incentive | Control (Education)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/11
Other Adverse Events (participants affected / at risk) | 0/22 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT02880176/Prot_SAP_000.pdf